CLINICAL TRIAL: NCT00690365
Title: A Non-interventional, Open Label, Phase IV Observational Study for the Safety and Efficacy of Switching to Quetiapine (Seroquel) in Outpatients With Schizophrenia Who Have Been Unsuccessfully Treated With Other Antipsychotics
Brief Title: Safety and Efficacy of Switching to Quetiapine in Outpatients With Schizophrenia
Acronym: Q-chase
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Panagiotis Pontikis, MD, Medical & Regulatory Affairs Director, AstraZeneca Greece, AstraZeneca S.A., Greece
Other Study IDs: NIS-NGR-SER-2007/1
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia
Keywords: Switching; Quetiapine; schizophrenia; unsuccessfully treated; antipsychotics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single-arm, phase IV, open-label, prospective, non interventional study in approximately 600 patients that will be followed for 6 months in order to evaluate the safety and efficacy of quetiapine. Patients will be switched over a 4 to 7 day cross-titration period from their previous antipsychotic medication to quetiapine according to the approved SPC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia at least 1 year prior to screening
* Inadequate response or poor safety /tolerability or non-compliance to previous antipsychotic medication
* Provision of Informed Consent prior to enrolment

Exclusion Criteria:

* Known hypersensitivity to active substance of excipients
* Patients receiving P450 3A4 inhibitors
* Pregnancy or lactation
* Substance abuse or dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety of quetiapine assessed through analysis of AE/SAE data (rate of patients presenting SAEs, rate of patients who discontinue treatment due to any AE, time to treatment discontinuation due to any AEs) | 5 visits (Day 0, Week 1, Week 4, Week 12, Week 24); SAEs will be reported during all study period

SECONDARY OUTCOMES:
Changes in the Clinical Global Impression of Severity and Improvement (CGI-S, CGI-I) and in Brief psychiatric Rating Scale (BPRS) from baseline to end of study treatment | 5 visits (Day 0, Week 1, Week 4, Week 12, Week 24)
Percentage of extra-pyramidal side effects assessed using the Simpson-Angus Scale (SAS) | Changes from baseline to end of study treatment or (6 months) or early withdrawal